CLINICAL TRIAL: NCT01605396
Title: A Phase II Randomized Trial of the Combination of Ridaforolimus and Exemestane, Compared to Ridaforolimus, Dalotuzumab and Exemestane in High Proliferation, Estrogen Receptor Positive Breast Cancer Patients
Brief Title: A Phase II Trial of Ridaforolimus and Exemestane, Compared to Ridaforolimus, Dalotuzumab and Exemestane in Participants With Breast Cancer (MK-8669-064)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8669-064; 2012-000335-11 (EudraCT Number); MK-8669-064 (Other: Merck)
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — ridaforolimus; dalotuzumab; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ridaforolimus + Dalotuzumab + Exemestane (Experimental): Participants receive ridaforolimus 10 mg orally (PO) every 5 days (QD x 5) plus dalotuzumab 10 mg/kg intravenously (IV) every week (QW) plus exemestane 25 mg PO every day (QD) in 28-day cycles until documented disease progression or unacceptable toxicity.
  Interventions: Drug: Ridaforolimus; Drug: Dalotuzumab; Drug: Exemestane
- Ridaforolimus + Exemestane (Active Comparator): Participants receive ridaforolimus 30 mg PO QD x 5 plus exemestane 25 mg PO QD treatment in 28-day cycles until documented disease progression or unacceptable toxicity.
  Interventions: Drug: Ridaforolimus; Drug: Exemestane

INTERVENTIONS:
Drug: Ridaforolimus — Ridaforolimus 10 mg tablet, administered PO at a dose of 10 mg (triplet) or 30 mg (doublet) depending upon randomization, on Days 1-5, 8-12, 15-19, & 22-26 of 28-day cycle.
  Other Names: MK-8669; AP23573
Drug: Dalotuzumab — Dalotuzumab administered 10 mg/kg IV weekly on Days 1, 8, 15, and 22 of 28-day cycle.
  Other Names: MK-0646; h7C10
  Arms: Ridaforolimus + Dalotuzumab + Exemestane
Drug: Exemestane — Exemestane 25 mg tablet administered PO QD.
  Other Names: Aromasin

SUMMARY:
The purpose of the study is to evaluate the efficacy of the triplet of ridaforolimus, dalotuzumab and exemestane compared to the combination of ridaforolimus and exemestane in post-menopausal participants with breast cancer. The primary hypothesis of the study is that the triplet of ridaforolimus, dalotuzumab and exemestane will improve progression free survival (PFS) compared to ridaforolimus and exemestane.

ELIGIBILITY:
Inclusion Criteria:

* Females with a histologically confirmed diagnosis of breast cancer that is metastatic or locally advanced (locally advanced tumors must not be amenable to

surgery or radiation therapy with curative intent) with the following pathological characteristics determined locally: estrogen receptor positive and Human Epidermal Growth Factor Receptor 2 (HER-2) negative, and Ki67 (a tumor marker) ≥ 15% determined by the central study laboratory

* Post-menopausal
* With advanced breast cancer whose disease was refractory to previous letrozole or anastrozole
* Has at least one confirmed measurable metastatic lesion
* Has a performance status ≤ 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Has a life expectancy of at least 3 months
* Adequate organ function

Exclusion Criteria:

* Is receiving any other concurrent systemic tumor therapy, including

hormonal agents and HER-2 inhibitors

* Previously received rapamycin or rapamycin analogs, including

ridaforolimus, temsirolimus, or everolimus

* Received prior treatment with Insulin-like Growth Factor 1 Receptor (IGF-1R) inhibitors, Phosphatidylinositol 3-Kinase (PI3K) inhibitors, or

other experimental agents that target PI3K, Protein Kinase B (AKT), or Mammalian Target of Rapamycin (mTOR) pathway

* Is receiving chronic corticosteroids administered at doses greater than

those used for normal replacement therapy

* Has active brain metastasis or leptomeningeal carcinomatosis; patients

with adequately treated brain metastases are eligible if they meet certain criteria

* Known allergy to macrolide antibiotics
* Has an active infection requiring antibiotics
* Significant or uncontrolled cardiovascular disease
* Poorly controlled Type 1 or 2 diabetes
* Is known to be Human Immunodeficiency Virus (HIV) positive
* Has a known history of active hepatitis B or C. Healthy carriers of hepatitis B are not allowed on this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-07-04 (Actual); Primary Completion 2014-02-19 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rugo HS, Tredan O, Ro J, Morales SM, Campone M, Musolino A, Afonso N, Ferreira M, Park KH, Cortes J, Tan AR, Blum JL, Eaton L, Gause CK, Wang Z, Im E, Mauro DJ, Jones MB, Denker A, Baselga J. A randomized phase II trial of ridaforolimus, dalotuzumab, and exemestane compared with ridaforolimus and exemestane in patients with advanced breast cancer. Breast Cancer Res Treat. 2017 Oct;165(3):601-609. doi: 10.1007/s10549-017-4375-5. Epub 2017 Jul 5. PMID 28681171

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 196 screened participants, 80 were randomized to either ridaforolimus plus dalotuzumab plus exemestane or ridaforolimus plus exemestane.
Groups:
- Ridaforolimus + Dalotuzumab + Exemestane: Participants received ridaforolimus 10 mg orally (PO) every 5 days (QD x 5) plus dalotuzumab 10 mg/kg intravenously (IV) every week (QW) plus exemestane 25 mg PO every day (QD) in 28-day cycles until documented disease progression or unacceptable toxicity.
- Ridaforolimus + Exemestane: Participants received ridaforolimus 30 mg PO QD x 5 plus exemestane 25 mg PO QD treatment in 28-day cycles until documented disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Ridaforolimus + Dalotuzumab + Exemestane | Ridaforolimus + Exemestane
Started | 40 | 40
Treated | 39 | 40
Completed | 0 | 0
Not Completed | 40 | 40
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-Compliance With Study Drug | 1 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Progressive Disease | 23 | 27
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Transfer Off Study | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ridaforolimus + Dalotuzumab + Exemestane | Ridaforolimus + Exemestane | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (9.0) | 57.7 (11.8) | 59.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 35 | 34 | 69
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 14 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 26 | 24 | 50
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 1. Progression-free Survival (PFS) According to Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Based on Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization to progressive disease, or death, whichever occurs first. Response was assessed according to RECIST 1.1 by BICR. According to RECIST 1.1, progressive disease (PD) was defined as a 20% relative increase in the sum of diameters (SOD) of target lesions, taking as reference the nadir SOD and an absolute increase of >5 mm in the SOD, or the appearance of new lesions. PFS was analyzed using the Kaplan-Meier method and median PFS (95% confidence interval [CI]) in weeks was reported for each treatment arm. Per protocol, participants remained on assigned treatment until disease progression. Participants who discontinued study treatment for reasons other than disease progression continued to be assessed by imaging until objective documentation of progression. All participants (including participants who discontinued study treatment) were followed for survival until investigator notification to discontinue.
Time Frame: From Day 1 through last post-study efficacy follow-up (up to ~19 months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ridaforolimus + Dalotuzumab + Exemestane | Ridaforolimus + Exemestane
Number analyzed (Participants) | 40 | 40
Weeks | 23.29 [8.71 to 38.43] | 31.86 [16.00 to 39.29]
Statistical Analysis 1: Comparison: Ridaforolimus + Dalotuzumab + Exemestane vs Ridaforolimus + Exemestane; Hazard ratio (HR) and p-value for treatment difference based on Cox regression model with Efron tie handling for treatment comparison (Ridaforolimus + Dalotuzumab + Exemestane arm versus Ridaforolimus + Exemestane arm); Test type: Superiority; p = 0.565, Regression, Cox; Hazard Ratio (HR) = 1.18, 80% CI 2-sided [0.81 to 1.72]

2. Secondary Outcome: Percent Change From Baseline in Sum of Target Lesion Diameters at Week 16
Description: The percent change from baseline to Week 16 in the sum of target lesion diameters as determined by anatomic imaging was defined as the line length (i.e., diameter) for each target lesion identified at baseline summed across all lesions at baseline, and separately at each post-baseline time point. The primary analysis was conducted using a constrained longitudinal data analysis (cLDA) method and target lesion measurements according to the BICR. Percent change from baseline in sum of target lesion diameters at Week 16 was reported for each treatment arm.
Time Frame: Baseline, Week 16
Population: All randomized participants with available Week 16 target lesion measurements.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ridaforolimus + Dalotuzumab + Exemestane | Ridaforolimus + Exemestane
Number analyzed (Participants) | 15 | 32
percent change | -19.3 (20.4) | -10.7 (28.5)

3. Secondary Outcome: 3. Percentage of Participants With Objective Response (Objective Response Rate [ORR]) According to Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Based on Blinded Independent Central Review (BICR).
Description: ORR was defined as the percentage of participants whose best response was complete response (CR; disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal) or partial response (PR; at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD) according to RECIST 1.1 and based on BICR. ORR was reported for each treatment arm. Per protocol, participants remained on assigned treatment until disease progression. Participants who discontinued study treatment for reasons other than disease progression continued to be assessed by imaging until objective documentation of progression.
Time Frame: From Day 1 through last post-study efficacy follow-up (up to ~19 months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ridaforolimus + Dalotuzumab + Exemestane | Ridaforolimus + Exemestane
Number analyzed (Participants) | 40 | 40
Percentage of Participants | 15.0 [5.7 to 29.8] | 25.0 [12.7 to 41.2]
Statistical Analysis 1: Comparison: Ridaforolimus + Dalotuzumab + Exemestane vs Ridaforolimus + Exemestane; Miettinen and Nurminen's method was used to compare ORR between the two treatment arms (Ridaforolimus + Dalotuzumab + Exemestane arm versus Ridaforolimus + Exemestane arm), and to calculate a p-value and 95% confidence interval (CI) for the difference in response rates; Test type: Other; p = 0.267, Miettinen and Nurminen's Method; Difference of Percentages = -10.0, 95% CI 2-sided [-27.8 to 8.0]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of analysis were censored at the date last known to be alive. OS was analyzed using the Kaplan-Meier method and median OS (95% confidence interval [CI]) in weeks was reported for each treatment arm. Per protocol, all participants (including participants who discontinued study treatment) were followed for survival until investigator notification to discontinue.
Time Frame: From Day 1 through last post-study efficacy follow-up (up to ~19 months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ridaforolimus + Dalotuzumab + Exemestane | Ridaforolimus + Exemestane
Number analyzed (Participants) | 40 | 40
Weeks | NA [NA to NA] — Median OS could not be calculated due to an insufficient number of deaths on study (i.e. median OS was not reached). | NA [60.6 to NA] — Median OS could not be calculated due to an insufficient number of deaths on study (i.e. median OS was not reached).
Statistical Analysis 1: Comparison: Ridaforolimus + Dalotuzumab + Exemestane vs Ridaforolimus + Exemestane; HR and p-value for treatment difference based on Cox regression model with Efron tie handling for treatment comparison (Ridaforolimus + Dalotuzumab + Exemestane arm versus Ridaforolimus + Exemestane arm); Test type: Other; p = 0.562, Regression, Cox; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [0.46 to 4.13]

ADVERSE EVENTS:
Time Frame: From Day 1 through Post Treatment visit at 4 weeks after last dose of treatment (up to ~17 months)
Description: All randomized participants who received at least one dose of study treatment. For nine participants who continued to receive treatment under compassionate use after database lock, safety data was not included in any study database but was reported to global safety.
Arm/Group | Ridaforolimus + Dalotuzumab + Exemestane | Ridaforolimus + Exemestane
All-Cause Mortality (participants affected / at risk) | 1/39 | 2/40
Serious Adverse Events (participants affected / at risk) | 8/39 | 17/40
Other Adverse Events (participants affected / at risk) | 39/39 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ridaforolimus + Dalotuzumab + Exemestane (N=39) | Ridaforolimus + Exemestane (N=40)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Oesophagitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ridaforolimus + Dalotuzumab + Exemestane (N=39) | Ridaforolimus + Exemestane (N=40)
Anaemia (Blood and lymphatic system disorders) | 6 (8) | 9 (11)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (5)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 3 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 4 (7)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (7) | 8 (11)
Diarrhoea (Gastrointestinal disorders) | 14 (31) | 15 (28)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (18) | 9 (11)
Oral pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 30 (54) | 36 (88)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (4)
Vomiting (Gastrointestinal disorders) | 8 (20) | 8 (8)
Asthenia (General disorders) | 10 (13) | 14 (15)
Chest pain (General disorders) | 0 (0) | 3 (4)
Chills (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 11 (13) | 7 (9)
Local swelling (General disorders) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 3 (6) | 10 (12)
Pyrexia (General disorders) | 4 (7) | 5 (5)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 4 (4) | 0 (0)
Gingivitis (Infections and infestations) | 2 (2) | 2 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (4) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 6 (6)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 6 (9) | 3 (3)
Blood cholesterol increased (Investigations) | 2 (2) | 4 (5)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3)
Platelet count decreased (Investigations) | 1 (1) | 5 (5)
Weight decreased (Investigations) | 3 (3) | 6 (6)
White blood cell count decreased (Investigations) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 15 (16) | 11 (13)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (14) | 10 (20)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (8)
Dizziness (Nervous system disorders) | 1 (1) | 6 (7)
Dysgeusia (Nervous system disorders) | 14 (16) | 6 (6)
Headache (Nervous system disorders) | 6 (6) | 13 (18)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 2 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 10 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 4 (7)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Onycholysis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 8 (12) | 8 (13)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 4 (5)
Lymphoedema (Vascular disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.